CLINICAL TRIAL: NCT07259304
Title: Social Health, Activity Behaviors, and Quality of Life Among Young Adult Cancer Survivors: A Longitudinal Study
Brief Title: Social Health, Activity Behaviors, and Quality of Life Among Young Adult Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-20-10; NCI-2021-05723 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-20-10 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); R37CA256867 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Central Nervous System Neoplasm; Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage IIA Cutaneous Melanoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; Hodgkin Lymphoma; Malignant Bone Neoplasm; Malignant Brain Neoplasm; Malignant Solid Neoplasm; Malignant Testicular Neoplasm; Non-Hodgkin Lymphoma; Pathologic Stage I Cutaneous Melanoma AJCC v8; Pathologic Stage IA Cutaneous Melanoma AJCC v8; Pathologic Stage IB Cutaneous Melanoma AJCC v8; Pathologic Stage II Cutaneous Melanoma AJCC v8; Pathologic Stage IIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIC Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage I Cervical Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Differentiated Thyroid Gland Carcinoma AJCC v8; Stage I Ovarian Cancer AJCC v8; Stage I Thyroid Gland Medullary Carcinoma AJCC v8; Stage I Uterine Corpus Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA Ovarian Cancer AJCC v8; Stage IA Uterine Corpus Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB Cervical Cancer AJCC v8; Stage IB Ovarian Cancer AJCC v8; Stage IB Uterine Corpus Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer AJCC v8; Stage IC Ovarian Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Differentiated Thyroid Gland Carcinoma AJCC v8; Stage II Ovarian Cancer AJCC v8; Stage II Thyroid Gland Medullary Carcinoma AJCC v8; Stage II Uterine Corpus Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIA Ovarian Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIB Ovarian Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Differentiated Thyroid Gland Carcinoma AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Thyroid Gland Medullary Carcinoma AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8
MeSH Terms: conditions — Central Nervous System Neoplasms; Hodgkin Disease; Bone Neoplasms; Brain Neoplasms; Testicular Neoplasms; Lymphoma, Non-Hodgkin; Uterine Cervical Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (actigraph, surveys): Patients complete surveys and wear an actigraph GT3X-BT accelerometer continuously for 7 days at baseline, 3, 6, and 12 months.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Other: Medical Device Usage and Evaluation — Wear an actigraph GT3X-BT accelerometer
Other: Quality-of-Life Assessment — Complete survey
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete survey

SUMMARY:
This study assesses how personal relationships (such as friendships, family relationships, or romantic partners) influence the physical activity (exercise) and well-being of young adult cancer survivors. Researchers also hope to learn how social relationships change after a cancer diagnosis, and how these changes might impact important health behaviors. The information provided may help researchers learn more about better ways to support young cancer patients in the future through interventions that help maintain good social relationships and health levels of physical activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize the trajectories of social health in young adult (YA) cancer patients.

II. Investigate the longitudinal associations between social health and activity behaviors in YA cancer patients.

III. Explore the effects of sociodemographic and clinical characteristics on the relationship between social health, activity behaviors, and quality of life.

OUTLINE:

Patients complete surveys over 40 minutes and wear an actigraph GT3X-BT accelerometer continuously for 7 days at baseline, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and/or treated with cancer between ages 18-39 at USC hospitals.
* Cancer types prototypical for adolescents and young adults (AYAs) and cancer stages I-III; select patients with stage IV disease may be eligible, with approval by the principal investigator (PI) and in consultation with the treating clinician.
* Must be within three months of a de novo cancer diagnosis at recruitment and on/indicated for curative therapy (any modality). Patients may continue on adjuvant therapy throughout duration of the study.
* Patients must have anticipated survival of >1-year at time of diagnosis.

Exclusion Criteria:

* Diagnosis of blood malignancies such as leukemias (these cancers have divergent treatment patterns of longer duration than other cancers and are more commonly pediatric cancers). Some early stage lymphomas with favorable prognoses may be eligible, with approval by the PI and in consultation with the treating clinician.
* Primary language other than English or Spanish.
* Inability to complete a survey and/or wear an accelerometer either per the patient or in consultation with the clinician's judgment.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed and/or treated with cancer between ages 18-39 at University of Southern California (USC) hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in trajectories of social health | Baseline up to 1 year
  Social health variables include the number, frequency and duration of hospitalizations, specifics of cancer diagnosis (i.e., stage at diagnosis, pertinent histology, recurrence or progression of disease), chemotherapy type, surgery related to cancer diagnosis, radiation field, immunotherapy type, and other relevant therapies related to cancer treatment.
  Changes in above variables will be measured using latent growth curve models to measure latent intercept (initial level), and the latent slope (rate of change) of social health variables during the course of therapy.
Rate of Change in trajectories of physical activity | Baseline up to 1 year
  Changes will be measured using latent growth curve models to measure latent intercept (initial level) and the latent slope (rate of change) of physical activity during the course of therapy.
Rate of Change in trajectories of quality of life | Baseline up to 1 year
  Changes will be measured using latent growth curve models to measure latent intercept (initial level) and the latent slope (rate of change) of quality of life during the course of therapy.
Moderation by gender | Up to 1 year
  Will conduct multi-group analyses by the categories of study moderators (e.g., gender, race/ethnicity, socioeconomic status [SES], health status). The strengths of group-specific pathways to link social health and activity behaviors to quality of life will be compared using the chi-square (χ2) difference test of model fit. The log-likelihood values with (versus [vs.] without) the equality constraints on the group-specific pathways to determine if the strength of associations estimated in the models significantly differ by the groups of each moderator (e.g., gender: female vs. male).
Moderation effect of race/ethnicity | Up to 1 year
  Moderation effect is analyzed by the interaction between the independent variable (X), and the moderator variable (Y) in a regression model, where the endpoint is the dependent variable (Z). Moderation effect is the endpoint itself, indicated by the significance of the interaction term's regression coefficient (B3), which shows how the relationship between X and Y changes depending on the level of Z. 'X' is social health, physical activity, and quality of life. 'Y' is race/ethnicity. 'Z' is moderation effect. The strengths of group-specific pathways to link social health and activity behaviors to quality of life will be compared using the chi-square (χ2) difference test of model fit.
Moderation effect of Socio-Economic Status (SES) | Up to 1 year
  Moderation effect is analyzed by the interaction between the independent variable (X), and the moderator variable (Y) in a regression model, where the endpoint is the dependent variable (Z). Moderation effect is the endpoint itself, indicated by the significance of the interaction term's regression coefficient (B3), which shows how the relationship between X and Y changes depending on the level of Z. 'X' is social health, physical activity, and quality of life. 'Y' is socio-economic status. 'Z' is moderation effect. The strengths of group-specific pathways to link social health and activity behaviors to quality of life will be compared using the chi-square (χ2) difference test of model fit.
Moderation effect of health status | Up to 1 year
  Moderation effect is analyzed by the interaction between the independent variable (X), and the moderator variable (Y) in a regression model, where the endpoint is the dependent variable (Z). Moderation effect is the endpoint itself, indicated by the significance of the interaction term's regression coefficient (B3), which shows how the relationship between X and Y changes depending on the level of Z. 'X' is social health, physical activity, and quality of life. 'Y' is health status. 'Z' is moderation effect. The strengths of group-specific pathways to link social health and activity behaviors to quality of life will be compared using the chi-square (χ2) difference test of model fit.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Miller, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States